CLINICAL TRIAL: NCT05003986
Title: A Phase 2, Open-Label, Single-Arm, Cohort Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of Sparsentan Treatment in Pediatric Subjects With Selected Proteinuric Glomerular Diseases
Brief Title: Study of Sparsentan Treatment in Pediatrics With Proteinuric Glomerular Diseases
Acronym: EPPIK
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Travere Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTRX-RE021-201
Record Dates: First submitted 2021-07-29; First posted 2021-08-13 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Focal Segmental Glomerulosclerosis; Minimal Change Disease; Immunoglobulin A Nephropathy; IgA Vasculitis; Alport Syndrome
Keywords: Alport, AS, FSGS, IgAN, IgAV, MCD, pediatrics, peds
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental; Nephrosis, Lipoid; Glomerulonephritis, IGA; IgA Vasculitis; Nephritis, Hereditary; Macular dystrophy, corneal type 1 | interventions — sparsentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Population 1: FSGS and/or MCD (Experimental): Subjects with selected proteinuric glomerular diseases associated with FSGS and MCD histological patterns
  Interventions: Drug: Sparsentan
- Population 2: IgAN, IgAV, or AS (Experimental): Subjects with kidney biopsy-confirmed immunoglobulin A nephropathy (IgAN), immunoglobulin A vasculitis (IgAV), or Alport syndrome (AS)
  Interventions: Drug: Sparsentan
- Population 3: IgAN (Experimental): Subjects with kidney biopsy-confirmed IgAN
  Interventions: Drug: Sparsentan

INTERVENTIONS:
Drug: Sparsentan — Population 1: 800 mg Sparsentan (oral suspension)
  Other Names: RE-021
  Arms: Population 1: FSGS and/or MCD
Drug: Sparsentan — Population 2: 400 mg Sparsentan (oral suspension)
  Other Names: RE-021
  Arms: Population 2: IgAN, IgAV, or AS
Drug: Sparsentan — Population 3: 400 mg Sparsentan (tablets)
  Other Names: RE-021
  Arms: Population 3: IgAN

SUMMARY:
To evaluate the safety, efficacy and tolerability of sparsentan oral suspension and tablets, and assess changes in proteinuria after once-daily dosing over 108 weeks.

DETAILED DESCRIPTION:
This is a multicenter, open-label, 112-week study of sparsentan in approximately 67 pediatric subjects aged ≥1 year to <18 years with selected proteinuric glomerular diseases, divided into 3 populations, defined as follows:

* Population 1: Subjects with selected proteinuric glomerular diseases associated with Focal Segmental Glomerulosclerosis (FSGS) and Minimal Change Disease (MCD) histological patterns
* Population 2: Subjects with kidney biopsy-confirmed immunoglobulin A nephropathy (IgAN), immunoglobulin A vasculitis (IgAV), or Alport syndrome (AS)
* Population 3: Subjects with kidney biopsy-confirmed IgAN

The study will evaluate long-term safety, tolerability, and efficacy with pharmacokinetic (PK) evaluations at Day 1 (Baseline), Day 2 (Visit 4), and Week 12 (Visit 9) in Population 1 and Population 2. In Population 3, PK values will be evaluated at Day 1 (Baseline) and at Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, and 96. For Population 1 and Population 2, subjects will be enrolled in 3 cohorts based on age ranges. For Population 3, subjects will be enrolled in one cohort.

Study Enrollment:

* Population 1: FSGS and/or MCD (30 subjects total)

  1. Cohort 1 (6 subjects): ≥8 years to <18 years
  2. Cohort 2 (18 subjects): ≥3 years to <8 years
  3. Cohort 3 (6 subjects): ≥1 year to <3 years
* Population 2: IgAN, IgAV, or AS (27 subjects total)

  1. Cohort 1 (9 subjects): ≥8 years to <18 years
  2. Cohort 2 (12 subjects): ≥5 years to <8 years
  3. Cohort 3 (6 subjects): ≥2 years to <5 years
* Population 3: IgAN (10 subjects total) 1. 10 subjects: ≥8 years to <18 years

ELIGIBILITY:
Inclusion Criteria for All Subjects (All Three Populations):

A subject must meet all of the following criteria to be eligible for participation in this study:

* The subject or parent/legal guardian (as appropriate) is willing and able to provide signed informed consent/assent, and where required, the subject is willing to provide assent before any screening procedures per local requirements.
* The subject has an estimated glomerular filtration rate (eGFR) ≥30 mL/min/1.73 m2 at screening.
* The subject has a mean seated blood pressure between the 5th and 95th percentile for sex and height.

Inclusion Criteria for Population 1:

* The subject is male or female ≥1 year at screening and <18 years of age at Day 1 (Baseline).
* The subject has a UP/C ≥1.5 g/g (170 mg/mmol) at screening AND one of the following:
* Kidney biopsy-proven FSGS or MCD histological patterns and clinical presentation consistent with primary FSGS or MCD and qualifying proteinuria at screening despite history or ongoing treatment with corticosteroids and/or other immunosuppressive disease-modifying agents.
* Documentation of a genetic mutation in a podocyte protein associated with FSGS or MCD. Subjects with a documented podocytic mutation do not require kidney biopsy.
* Kidney biopsy-proven FSGS histological pattern with medical history and clinical presentation consistent with maladaptive cause of the lesion.

Note: The kidney biopsy may have been performed at any time in the past but must include light microscopy and electron microscopy characteristics and/or immunofluorescence findings consistent with FSGS or MCD.

Inclusion Criteria for Population 2:

* The subject is male or female ≥2 years at screening and <18 years of age at Day 1 (Baseline).
* The subject has UP/C ≥0.6 g/g (68 mg/mmol) at screening AND one of the following diagnoses:
* Kidney biopsy-confirmed IgAN, IgAV, or AS
* Diagnosis of AS by genetic testing (pathogenic X-linked Collagen, Type IV, Alpha-5 (COL4A5) mutation OR autosomal-recessive mutations in both alleles of Collagen, Type IV, Alpha-3 (COL4A3) and/or Collagen, Type IV, Alpha-4 (COL4A4) OR autosomal-dominant COL4A3 and/or COL4A4 and digenic mutations [ie, simultaneous mutations in 2 of the COL4A3, COL4A4, and COL4A5 genes])

Inclusion Criteria for Population 3:

* The subject is male or female ≥8 years at screening and <18 years of age at Day 1 (Baseline).
* The subject has UP/C ≥1.0 g/g (113 mg/mmol) at screening AND has kidney biopsy-confirmed IgAN
* Subject weighs ≥40 kg
* The subject has been on ACEI and/or ARB therapy for at least 12 weeks prior to screening

Exclusion Criteria for All Subjects (All Three Populations):

A subject who meets any of the following will be excluded from this study:

* The subject weighs <7.3 kg at screening.
* The subject has FSGS or MCD histological pattern secondary to viral infections, drug toxicities, or malignancies.
* The subject has immunoglobulin A (IgA) glomerular deposits not in the context of primary IgAN or IgAV (ie, secondary to another condition; eg, systemic lupus erythematosus and liver cirrhosis).
* The subject has had an acute onset or presentation of glomerular disease or a diagnostic biopsy or a relapse of glomerular disease requiring new or different class of immunosuppressive treatment (including, but not limited to, systemic corticosteroids, calcineurin inhibitors and mycophenolate mofetil, abatacept, cyclophosphamide, rituximab, ofatumumab, and ocrelizumab) within 6 months before screening.
* Subjects taking chronic immunosuppressive medications (including systemic steroids) not on a stable dose for ≥1 month before screening.
* The subject requires any of the prohibited concomitant medications as defined in the study protocol.
* The subject has undergone any organ transplantation, with the exception of corneal transplants.
* The subject has a documented history of congenital or acquired heart failure (modified Ross heart failure classification for children Class II to Class IV) and/or previous hospitalization for heart failure or unexplained dyspnea, orthopnea, paroxysmal nocturnal dyspnea, ascites, and/or peripheral edema.
* The subject has hemodynamically significant cardiac valvular disease.
* The subject has clinically significant congenital vascular disease.
* The subject has jaundice, hepatitis, or known hepatobiliary disease, or alanine aminotransferase and/or aspartate aminotransferase >2 times the upper limit of the normal range at screening.
* The subject has a history of malignancy within the past 2 years.
* The subject has a screening hematocrit <27% (0.27 L/L) or a hemoglobin value <9 g/dL (90 g/L).
* The subject has a screening potassium value >5.5 milliequivalent (mEq)/L (5.5 mmol/L).
* The subject has any abnormal clinical laboratory screening values that are considered by the Investigator to be clinically significant.
* The subject has a history of allergic response to any angiotensin II antagonist or endothelin receptor antagonist, including sparsentan, or has a hypersensitivity to any of the excipients in the study medication.
* The female subject is pregnant, plans to become pregnant during the course of the study, or is breastfeeding.
* Female subjects of childbearing potential, beginning at menarche, who do not agree to use 1 highly reliable (ie, can achieve a failure rate of <1% per year) method of contraception from 7 days before the first dose of the study medication until 28 days after the last dose of study medication. Examples of highly reliable contraception methods include stable oral, implanted, transdermal, or injected contraceptive hormones associated with the inhibition of ovulation or an intrauterine device. One additional barrier method must also be used during vaginal sexual activity, such as a diaphragm, diaphragm with spermicide (preferred), or male partner's use of male condom or male condom with spermicide (preferred), from Day 1/Randomization until 28 days after the last dose of study medication. Female subjects of childbearing potential are defined as those who are fertile after menarche, unless permanently sterile; permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy. All female subjects of childbearing potential must have a negative serum pregnancy test result at screening (Visit 1) and a negative urine pregnancy test result, with positive results confirmed by serum, at every study visit from Day 1 (Visit 3) and after.

Note: Before menarche, pregnancy testing and contraceptive use are not required. However, subjects and their parents/legal guardians must be advised that, immediately upon menarche, subjects will be required to begin pregnancy testing and initiate contraceptive use. This requirement cannot be waived.

* The subject has participated in a study of another study medication within 28 days before screening or plans to participate in such a study during the course of this study.
* The subject has had prior exposure to sparsentan.
* The subject or parent/legal guardian (as appropriate), in the opinion of the Investigator, are unable to adhere to the requirements of the study including but not limited to, a history of noncompliance and/or any other reason that causes the Investigator to believe the subject would not be a good candidate for the study.
* For Population 3 - the subject is unable to swallow the study medication tablets whole.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 67 (Estimated)
Dates: Start 2021-08-12 (Actual); Primary Completion 2027-03-12 (Estimated); Study Completion 2027-04-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), AEs leading to treatment discontinuation, and adverse events of interest (AEOIs) | After the last patient has undergone the week 108 visit (Visit 15).
  The incidence of TEAEs, SAEs, AEs leading to treatment discontinuation, and AEOIs
Urine protein/creatinine ratio (UP/C) at week 108 | After the last patient has undergone the Week 108 visit (Visit 15)
  Change from baseline in UP/C over 108 weeks

SECONDARY OUTCOMES:
Observed plasma Pharmacokinetic (PK) concentrations | At scheduled Day 1, Day 2 and Week 12 visits for Population 1 and 2. At scheduled Day 1 and Week 4, 8, 12, 24, 36, 48, 60, 72, 84, and 96 visits for Population 3.
  Observed plasma PK concentrations at scheduled timepoints and visits
Steady-state PK parameters area under the plasma concentration-time curve during a dosing interval ([AUCτ]) | Week 108
  Steady-state PK parameters [AUCτ]
Steady-state PK parameters [Cmax_ss] | Week 108
  Maximum steady-state plasma drug concentration [Cmax_ss]
Steady-state PK parameters [Cmin_ss] | Week 108
  Minimum steady-state plasma drug concentration [Cmin_ss]
Urine albumin/creatinine ratio (UA/C) over 108 weeks | Week 108
  Change from baseline in UA/C over 108 weeks
Estimated glomerular filtration rate (eGFR) over 108 weeks | Week 108
  Change from baseline in eGFR over 108 weeks
Proportion of subjects achieving complete remission of proteinuria | Week 108
  The proportion of subjects achieving complete remission of proteinuria, defined as UP/C <0.3 g/g over 108 weeks
Proportion of subjects with FSGS and/or MCD histological patterns achieving partial remission | Week 108
  The proportion of subjects with FSGS and/or MCD histological patterns achieving partial remission defined as UP/C ≤1.5 g/g and >40% reduction in UP/C over 108 weeks
Proportion of subjects who discontinue study medication due to inability to tolerate the oral suspension | Week 108
  The proportion of subjects who discontinue study medication due to inability to tolerate the smell, taste, aftertaste, volume of administration, or method of administration of oral suspension in Population 1 and Population 2

CONTACTS AND LOCATIONS:
Overall Officials: Radko Komers, MD, PhD, Study Director — Travere Therapeutics, Inc.
Locations (47):
- United States (23):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Nemours Children's Hospital, Wilmington, Delaware
  - University of Miami, Leonard M. Miller School of Medicine, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - University of Iowa, Stead Family Children's Hospital, Iowa City, Iowa
  - Floating Hospital for Children at Tufts Medical Center, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota, Masonic Children's Hospital, Minneapolis, Minnesota
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Cohen Children's Medical Center, New Hyde Park, New York
  - Fink Children's Ambulatory Care Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Atrium Health Levine Children's Hospital, Charlotte, North Carolina
  - Duke Molecular Physiology Institute, Durham, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center (OUHSC), Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - UT Health - John P. and Kathrine G. McGovern Medical School, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Germany (3):
  - Uniklinik Köln, Klinik und Poliklinik für Kinder- und Jugendmedizin, Cologne
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Heidelberg - Angelika Lautenschläger - Kinderklinik, Heidelberg
- Italy (5):
  - Policlinico Bari Ospedale Pediatrico Giovanni XXIII, Bari
  - IRCCS Istituto Giannina Gaslini, Genova
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedale Università di Padova, Padua
  - Ospedale Pediatrico Bambino Gesù, Roma
- Netherlands (2):
  - Emma Kinderziekenhuis, Amsterdam
  - Radboud Universitair Medisch Centrum, Nijmegen
- Poland (3):
  - Uniwersytecki Szpital Dziecięcy w Krakowie, Krakow
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Instytut Pomnik - Centrum Zdrowia Dziecka, Warsaw
- Spain (4):
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
- Sweden (2):
  - Drottning Silvias Barn- och Ungdomssjukhus, Gothenburg
  - Karolinska Universitetssjukhuset Huddinge, Stockholm
- United Kingdom (5):
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol Royal Hospital for Children, Bristol
  - NHS Greater Glasgow and Clyde, Royal Hospital for Children, Glasgow
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London
  - Manchester University NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Requests for clinical trial data, including language stating its intended use, should be directed to datarequest@travere.com. If approved, the requested information will be provided to the requestor after signing a data access agreement. Requests can be made following completion of the study and full publication of the study data in a peer reviewed journal for up to 36 months following its publication. Travere reserves the right to decline or recommend modifications to a request if it does not comply with the data sharing policy or if it is determined that the request is made by a biased source.
Time Frame: Requests can be made following completion of the study and full publication of the study data in a peer reviewed journal for up to 36 months following its publication.
Access Criteria: Requires submission and approval of intended use and a data sharing agreement.
URL: http://datarequest@travere.com

REFERENCES:
- [Derived] Rheault MN. Treatment Approaches for Alport Syndrome. J Am Soc Nephrol. 2025 Sep 12;37(1):172-9. doi: 10.1681/ASN.0000000897. Online ahead of print. PMID 40938675
- See also: Sponsor Website — http://travere.com
- See also: Study Website — https://EPPIKclinicalstudy.com